CLINICAL TRIAL: NCT00999271
Title: On the Role of Glucose-dependent Insulinotropic Polypeptide, GIP, in Postprandial Metabolism in Humans
Brief Title: Glucose-dependent Insulinotropic Polypeptide (GIP) and Lipid Metabolism
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: University of Copenhagen, University of Copenhagen
Other Study IDs: HD-2009-0025
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Healthy Subjects
Keywords: Glucose-dependent insulinotropic polypeptide; gastric emptying; appetite; energy intake; lipid metabolism

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy subjects: 30 healthy subjects without family history of diabetes or gastrointestinal disease, a normal oral glucose tolerance test (OGTT) and no intake of medicine
  Interventions: Other: Incretin hormone - Glucose-dependent insulinotropic polypeptide (GIP)

INTERVENTIONS:
Other: Incretin hormone - Glucose-dependent insulinotropic polypeptide (GIP) — two different dosages:
  * 0.8 pmol/kg/min
  * 1.5 pmol/kg/min for 300 minutes

SUMMARY:
The aim of this proposal is to examine whether endogenous GIP and exogenous GIP alone and in combination with insulin affect gastric emptying (GE), appetite, energy intake, energy expenditure (EE) and plasma levels of triglycerides (TAG), free fatty acids FFA) and glycerol in man.

ELIGIBILITY:
Inclusion Criteria:

* Informed oral and written consent
* Caucasians over the age of 18 years
* Normal 75 g oral glucose tolerance test (OGTT)
* Normal blood haemoglobin concentration
* Normal plasma lipid profile

Exclusion Criteria:

* First-degree relatives with diabetes and familial hypertriglyceridemia

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark